CLINICAL TRIAL: NCT01560650
Title: Effect of the Intensity of Continuous Renal Replacement Therapy in Patients With Cardiac Surgery Associated Acute Kidney Injury (CRITERIA STUDY)
Brief Title: Effect of the Intensity of Continuous Renal Replacement Therapy in Patients With Acute Kidney Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wei Shi (Other)
Responsible Party: Sponsor-Investigator, Wei Shi, Director of renal division of Guangdong General Hospital, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LXL-CRRT2535
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Acute Kidney Injury
Keywords: CRRT; cardiac surgery associated acute kidney injury; Intensity
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose (35ml/kg/h) (Experimental): > = 18 years of age, CRRT indications for acute kidney injury (RIFLE criteria) patients with cardiac surgery, was given filtration at a rate of 35 mL/kg/h.
  Interventions: Device: CRRT
- low dose (25ml/kg/h) (Experimental): > = 18 years of age, CRRT indications for acute kidney injury (RIFLE criteria) patients with cardiac surgery, was given filtration at a rate of 25 mL/kg/h.
  Interventions: Device: CRRT

INTERVENTIONS:
Device: CRRT — Difference dose of CRRT

SUMMARY:
The current international Continuous Renal Replacement Therapy (CRRT) replacement fluid doses of 35 ml/kg/h is better, but the result is according to white people, black people . It is Whether the best amount of replacement fluid for Chinese people, it is unclear. Especially,there is little evidence about the optimal dose from randomized trials in Cardiac surgery associated acute kidney injury (CSA-AKI )required CRRT,According to the clinical situation, the design of replacement fluid to 25 ml/kg/h.The observation of two doses 14 days, 28 days, 90 days survival and renal function.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a major complication in patients with cardiac surgery and is an independent predictor of mortality. However, the optimal intensity of renal replacement therapy for such patients is still controversial. we randomly assigned the patients with Cardiac surgery-associated acute kidney injury (CSA-AKI) to continuous renal replacement therapy with different treatment dose (35ml / kg / h or 25ml/kg／h),The primary study outcome was death from any cause within 14, 28 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* > = 18 years of age, CRRT indications for acute kidney injury (RIFLE criteria) patients with cardiac surgery

Exclusion Criteria:

* < 18 years old,
* with chronic kidney disease,
* dialysis history, to leave the ICU patients with acute kidney injury (AKI). - chronic kidney disease,
* all causes kidney damage (pathology, hematuria, and radiographic abnormalities)> = 3 months or glomerular filtration rate < 60ml/min for 3 months or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2011-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
death from any cause | 14, 28 ,90 and 365 days after randomization
  The primary study outcome was death from any cause within 14, 28 ,90 and 365 days after randomization.

SECONDARY OUTCOMES:
renal outcome of survivors | 14, 28 ,90 and 365 days after randomization
  Secondary outcomes were renal outcome of survivors14, 28 ,90 and 365 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Nephrology Department,Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787